CLINICAL TRIAL: NCT02118428
Title: AIMS Study: African Investigation of Mirasol System for Whole Blood. Clinical and Biological Efficacy of Mirasol-treated Fresh Whole Blood for the Prevention of Transfusion-transmitted Malaria
Brief Title: Clinical and Biological Efficacy of Mirasol-treated Fresh Whole Blood for the Prevention of Transfusion-transmitted Malaria
Acronym: AIMS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Terumo BCTbio (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: CTS-5031
Record Dates: First submitted 2014-02-27; First posted 2014-04-21 (Estimated); Results first posted 2019-05-10 (Actual); Last update posted 2019-05-10 (Actual); Status verified 2019-02

CONDITIONS: Malaria
Keywords: whole blood; transfusion; Plasmodium; Malaria; Pathogen Reduction Technology; Whole blood transfusion
MeSH Terms: conditions — Malaria

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mirasol (Experimental): Transfusions with Mirasol-treated whole blood
  Interventions: Device: Mirasol-treated Whole Blood
- Control (Active Comparator): Transfusions with untreated whole blood
  Interventions: Biological: Untreated Whole Blood

INTERVENTIONS:
Device: Mirasol-treated Whole Blood — Transfusion with fresh Whole Blood treated with the Mirasol Pathogen Reduction Technology System for Whole Blood
  Arms: Mirasol
Biological: Untreated Whole Blood — Transfusion with untreated fresh Whole Blood
  Arms: Control

SUMMARY:
The trial will evaluate the efficacy of the Mirasol Pathogen Reduction Technology for Whole Blood to prevent Malaria transmission by transfusion of whole blood.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Patient is blood group O+
* Anticipated to be hospitalized for at least 3 consecutive days after initial study transfusion
* Expected to require no more than 2 units of Fresh Whole Blood in the 3 days following randomization
* Agree to return to the hospital for the follow-up visits
* Women of Child Bearing Potential must have a negative pregnancy test within 72 hours before randomization when warranted and must agree to practice a medically acceptable contraception regimen or agree to abstain from heterosexual intercourse during their study participation.
* Patient or legally authorized representative has given written informed consent

Exclusion Criteria:

* Symptoms of clinical malaria (confirmed by microscopy)
* Patient has received antimalarial treatment within 7 days prior to randomization
* Fever (Central body temperature greater than 38.5°C)
* Massive bleeding expected to require more than two Fresh Whole Blood units within 3 days from randomization
* Transfusion(s) of a blood product within 1 month prior to randomization
* Acute or chronic medical disorder that, in the opinion of the investigator, would impair the ability of the patient to receive protocol treatment
* Previous treatment with other pathogen-reduced blood products
* Females who are pregnant

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 227 (Actual)
Dates: Start 2014-03; Primary Completion 2014-12 (Actual); Study Completion 2014-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shirley Owusu-Ofori, MD, Principal Investigator — Komfo Anokye Teaching Hospital
Locations (1):
- Komfo Anokye Teaching Hospital, Kumasi, Ghana

REFERENCES:
- [Derived] Allain JP, Owusu-Ofori AK, Assennato SM, Marschner S, Goodrich RP, Owusu-Ofori S. Effect of Plasmodium inactivation in whole blood on the incidence of blood transfusion-transmitted malaria in endemic regions: the African Investigation of the Mirasol System (AIMS) randomised controlled trial. Lancet. 2016 Apr 23;387(10029):1753-61. doi: 10.1016/S0140-6736(16)00581-X. PMID 27116282

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 227 total were enrolled, but one participant was ineligible prior to randomization.
Groups:
- Control: Transfusions with untreated whole blood
  Untreated Whole Blood: Transfusion with fresh Whole Blood
- Unassigned: Enrolled subjects who became ineligible prior to randomization to either Mirasol or Control
Period: Overall Study
Arm/Group | Mirasol | Control | Unassigned
Started | 113 | 113 | 1
Received Study Transfusion | 111 | 112 | 0
Completed | 100 | 104 | 0
Not Completed | 13 | 9 | 1
Not completed — Physician Decision | 0 | 1 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 0
Not completed — Death | 7 | 5 | 0
Not completed — Lost to Follow-up | 3 | 1 | 0
Not completed — Screen Failure or Became Inelegible | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety population = all randomized subjects who underwent at least 1 study transfusion, independent of the outcome or successful completion of the procedure
Groups:
- Total: Total of all reporting groups
Arm/Group | Mirasol | Control | Total
Number analyzed (Participants) | 111 | 112 | 223
Age, Continuous [Mean (Standard Deviation); unit: years] | 38.9 (15.3) | 40.7 (17.0) | 39.8 (16.2)
Age, Customized [Count of Participants; unit: Participants]
  18-39 years | 62 | 67 | 129
  40-59 years | 35 | 28 | 63
  >=60 years | 14 | 17 | 31
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 77 | 84 | 161
  Male | 34 | 28 | 62
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 111 | 112 | 223
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Height [Mean (Standard Deviation); unit: meter] | 1.62 (0.08) | 1.63 (0.07) | 1.62 (0.08)
Weight [Mean (Standard Deviation); unit: kilogram] | 62.7 (13.4) | 63.9 (12.0) | 63.3 (12.7)
Body Mass Index [Mean (Standard Deviation); unit: kilogram/meter²] | 24.0 (4.9) | 24.2 (4.4) | 24.1 (4.6)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With Incidence of Transfusion-transmitted Malaria
Description: Percentage of Participants who contracted transfusion-transmitted malaria (TTM)
Time Frame: Up to 28 (+4) days after the initial whole blood transfusion (measured within 24 hours prior to each transfusion and at 24 (± 4) hours, 2 days, 3 days, 7 (+1) days, and 28 (+4) days after the initial whole blood transfusion)
Population: Evaluable population = randomized subjects who received up to 2 whole blood transfusions and no non-study blood products, who did not receive any anti-malarial treatment, who had no significant protocol deviations and who additionally were non parasitemic pre-transfusion and received at least one parasitemic fresh whole blood product
Measure: Number; unit: Percentage of participants
Arm/Group | Mirasol | Control
Number analyzed (Participants) | 28 | 37
Percentage of participants | 3.6 | 21.6

2. Secondary Outcome: Bacterial Contamination of Fresh Whole Blood (FWB) Products
Description: Bacterial culture on blood products - products were collected within 7 days before transfusion to the study subject.
  Control products were only sampled post-collection, so no results for post-Mirasol treatment.
  All samples in Mirasol group that were positive post-collection became negative post-Mirasol treatment.
  All samples in Mirasol group that were positive post-Mirasol treatment were negative post-collection. These samples were likely contaminated in the clinical laboratory after Mirasol treatment during sampling for culture.
Time Frame: immediately post-blood product collection & within 7 days before transfusion, post-Mirasol treatment (within 24 hours post-blood product collection) & within 7 days before transfusion
Population: Intent-to-treat = All randomized subjects who underwent at least 1 study transfusion
Measure: Number (95% Confidence Interval); unit: percentage of blood product samples
Arm/Group | Mirasol | Control
Number analyzed (Participants) | 111 | 112
percentage of blood product samples
  Positive post-collection | 3.3 [1.2 to 7.0] | 3.2 [1.2 to 6.9]
  Positive post-Mirasol treatment | 6.6 [3.5 to 11.3] | NA [NA to NA] — Control products are not Mirasol treated, so no post-Mirasol sample taken.

3. Secondary Outcome: Hematology Parameter in Fresh Whole Blood (FWB) Products - Hematocrit
Description: Hematocrit measurement in FWB products. Blood products were collected independently from study enrollment and stored for maximum of 7 days before assignment/transfusion to a study subject.
Time Frame: Post-blood product collection (Day -7 to Day 0 per transfusion), prior to transfusion (Day 0 per transfusion)
Population: Intent-to-treat = All randomized subjects who underwent at least 1 study transfusion
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Mirasol | Control
Number analyzed (Participants) | 111 | 112
percentage
  Hematocrit, post-collection | 38.14 (3.20) | 38.10 (3.03)
  Hematocrit, prior to transfusion | 35.54 (2.81) | 37.66 (2.77)

4. Secondary Outcome: Hematology Parameter in Fresh Whole Blood Products - Total Hemoglobin
Description: Total hemoglobin measurement in Fresh Whole Blood products. Blood products were collected independently from study enrollment and stored for maximum of 7 days before assignment/transfusion to a study subject.
Time Frame: Post-blood product collection (Day -7 to Day 0 per transfusion), prior to transfusion (Day 0 per transfusion)
Population: Intent-to-treat = All randomized subjects who underwent at least 1 study transfusion
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Mirasol | Control
Number analyzed (Participants) | 111 | 112
g/dL
  Total hemoglobin, post-collection | 12.98 (1.18) | 12.93 (1.13)
  Total hemoglobin, prior to transfusion | 11.97 (0.98) | 12.74 (1.03)

5. Secondary Outcome: Hematology Parameter in Fresh Whole Blood Products - Red Blood Cell (RBC) Count
Description: RBC count in Fresh Whole Blood products. Blood products were collected independently from study enrollment and stored for maximum of 7 days before assignment/transfusion to a study subject.
Time Frame: Post-blood product collection (Day -7 to Day 0 per transfusion), prior to transfusion (Day 0 per transfusion)
Population: Intent-to-treat = All randomized subjects who underwent at least 1 study transfusion
Measure: Mean (Standard Deviation); unit: Cells x 10e12/L
Arm/Group | Mirasol | Control
Number analyzed (Participants) | 111 | 112
Cells x 10e12/L
  RBC count, post-collection | 4.58 (0.49) | 4.57 (0.52)
  RBC count, prior to transfusion | 4.20 (0.49) | 4.47 (0.47)

6. Secondary Outcome: Hematology Parameter in Fresh Whole Blood Products - Platelet Count
Description: Platelet count in Fresh Whole Blood products. Blood products were collected independently from study enrollment and stored for maximum of 7 days before assignment/transfusion to a study subject.
Time Frame: Post-blood product collection (Day -7 to Day 0 per transfusion), prior to transfusion (Day 0 per transfusion)
Population: Intent-to-treat = All randomized subjects who underwent at least 1 study transfusion
Measure: Mean (Standard Deviation); unit: Cells x 10e9/L
Arm/Group | Mirasol | Control
Number analyzed (Participants) | 111 | 112
Cells x 10e9/L
  Platelet count, post-collection | 156.2 (44.3) | 156.9 (46.2)
  Platelet count, prior to transfusion | 85.3 (37.9) | 101.3 (57.2)

7. Secondary Outcome: Hematology Parameter in Fresh Whole Blood Products - White Blood Cell (WBC) Count
Description: WBC count in Fresh Whole Blood products. Blood products were collected independently from study enrollment and stored for maximum of 7 days before assignment/transfusion to a study subject.
Time Frame: Post-blood product collection (Day -7 to Day 0 per transfusion), prior to transfusion (Day 0 per transfusion)
Population: Intent-to-treat = All randomized subjects who underwent at least 1 study transfusion
Measure: Mean (Standard Deviation); unit: Cells x 10e9/L
Arm/Group | Mirasol | Control
Number analyzed (Participants) | 111 | 112
Cells x 10e9/L
  WBC, post-collection | 4.32 (1.05) | 4.45 (1.16)
  WBC, prior to transfusion | 3.69 (1.08) | 3.74 (1.39)

8. Secondary Outcome: Biochemistry Parameter in Fresh Whole Blood Products - Potassium
Description: Potassium measurement in Fresh Whole Blood products. Blood products were collected independently from study enrollment and stored for maximum of 7 days before assignment/transfusion to a study subject.
Time Frame: Post-blood product collection (Day -7 to Day 0 per transfusion), prior to transfusion (Day 0 per transfusion)
Population: Intent-to-treat = All randomized subjects who underwent at least 1 study transfusion
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Mirasol | Control
Number analyzed (Participants) | 111 | 112
mmol/L
  Potassium, post-collection | 3.61 (2.55) | 3.85 (3.33)
  Potassium, prior to transfusion | 14.97 (7.71) | 7.16 (3.27)

9. Secondary Outcome: Hematology Parameter in Patients - Hematocrit
Description: Hematocrit measure in study participants. Study participants may have received 1 or 2 blood product transfusions over 3 days while on study. These measurements were taken relative to the first transfusion only, for consistency.
Time Frame: Days 0, 1, 2, 3, 7, 28
Population: Intent-to-treat = All randomized subjects who underwent at least 1 study transfusion
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Mirasol | Control
Number analyzed (Participants) | 111 | 112
percentage
  Day 0 | 19.69 (5.40) | 19.52 (5.01)
  Day 1 | 24.25 (5.47) | 24.08 (4.21)
  Day 2 | 24.50 (4.48) | 25.48 (4.76)
  Day 3 | 24.72 (4.70) | 25.68 (4.77)
  Day 7 | 26.62 (4.88) | 26.92 (4.62)
  Day 28 | 28.61 (6.20) | 29.68 (5.56)

10. Secondary Outcome: Hematology Parameter in Patients - Total Hemoglobin
Description: Total hemoglobin measure in study participants. Study participants may have received 1 or 2 blood product transfusions over 3 days while on study. These measurements were taken relative to the first transfusion only, for consistency.
Time Frame: Days 0, 1, 2, 3, 7, 28
Population: Intent-to-treat = All randomized subjects who underwent at least 1 study transfusion
Measure: Mean (Standard Deviation); unit: g/dL
Arm/Group | Mirasol | Control
Number analyzed (Participants) | 111 | 112
g/dL
  Day 0 | 6.71 (1.97) | 6.71 (1.79)
  Day 1 | 8.53 (2.02) | 8.49 (1.55)
  Day 2 | 8.49 (1.58) | 8.83 (1.64)
  Day 3 | 8.57 (1.58) | 8.91 (1.65)
  Day 7 | 9.07 (1.75) | 9.18 (1.60)
  Day 28 | 9.72 (2.17) | 10.14 (1.9)

11. Secondary Outcome: Hematology Parameter in Patients - Platelet Count
Description: Platelet count in study participants. Study participants may have received 1 or 2 blood product transfusions over 3 days while on study. These measurements were taken relative to the first transfusion only, for consistency.
Time Frame: Days 0, 1, 2, 3, 7, 28
Population: Intent-to-treat = All randomized subjects who underwent at least 1 study transfusion
Measure: Mean (Standard Deviation); unit: Cells x 10e9/L
Arm/Group | Mirasol | Control
Number analyzed (Participants) | 111 | 112
Cells x 10e9/L
  Day 0 | 238.0 (168.79) | 234.50 (147.03)
  Day 1 | 202.40 (155.85) | 206.0 (121.47)
  Day 2 | 229.30 (145.56) | 228.20 (132.68)
  Day 3 | 235.50 (139.11) | 235.70 (124.79)
  Day 7 | 324.40 (152.79) | 332.40 (156.16)
  Day 28 | 269.10 (115.21) | 271.50 (126.15)

12. Secondary Outcome: Hematology Parameter in Patients - Red Blood Cell (RBC) Count
Description: RBC count in study participants. Study participants may have received 1 or 2 blood product transfusions over 3 days while on study. These measurements were taken relative to the first transfusion only, for consistency.
Time Frame: Days 0, 1, 2, 3, 7, 28
Population: Intent-to-treat = All randomized subjects who underwent at least 1 study transfusion
Measure: Mean (Standard Deviation); unit: Cells x 10e12/L
Arm/Group | Mirasol | Control
Number analyzed (Participants) | 111 | 112
Cells x 10e12/L
  Day 0 | 2.51 (0.75) | 2.52 (0.72)
  Day 1 | 3.05 (0.75) | 3.02 (0.60)
  Day 2 | 3.12 (0.66) | 3.27 (0.71)
  Day 3 | 3.15 (0.70) | 3.30 (0.73)
  Day 7 | 3.35 (0.70) | 3.41 (0.68)
  Day 28 | 3.60 (0.84) | 3.75 (0.72)

13. Secondary Outcome: Hematology Parameter in Patients - White Blood Cell (WBC) Count
Description: WBC count in study participants. Study participants may have received 1 or 2 blood product transfusions over 3 days while on study. These measurements were taken relative to the first transfusion only, for consistency.
Time Frame: Days 0, 1, 2, 3, 7, 28
Population: Intent-to-treat = All randomized subjects who underwent at least 1 study transfusion
Measure: Mean (Standard Deviation); unit: Cells x 10e9/L
Arm/Group | Mirasol | Control
Number analyzed (Participants) | 111 | 112
Cells x 10e9/L
  Day 0 | 10.34 (10.01) | 9.94 (6.97)
  Day 1 | 8.71 (5.64) | 8.07 (4.02)
  Day 2 | 7.91 (7.11) | 7.54 (4.80)
  Day 3 | 7.42 (6.42) | 7.09 (4.99)
  Day 7 | 7.15 (7.22) | 7.22 (4.96)
  Day 28 | 5.88 (5.0) | 5.48 (2.95)

14. Secondary Outcome: Biochemistry Parameter in Patients - Potassium
Description: Potassium measure in study participants. Study participants may have received 1 or 2 blood product transfusions over 3 days while on study. These measurements were taken relative to the first transfusion only, for consistency.
Time Frame: Days 0, 1, 2, 3
Population: Intent-to-treat = All randomized subjects who underwent at least 1 study transfusion
Measure: Mean (Standard Deviation); unit: mmol/L
Arm/Group | Mirasol | Control
Number analyzed (Participants) | 111 | 112
mmol/L
  Day 0 | 4.12 (0.85) | 4.17 (0.80)
  Day 1 | 4.14 (0.75) | 3.80 (0.49)
  Day 2 | 3.90 (0.69) | 3.97 (0.63)
  Day 3 | 4.00 (0.69) | 3.93 (0.61)

15. Secondary Outcome: Coagulation Parameter in Patients - Prothrombin Time
Description: Prothrombin time measure in study participants. Study participants may have received 1 or 2 blood product transfusions over 3 days while on study. These measurements were taken relative to the first transfusion only, for consistency.
Time Frame: Days 0, 1, 2, 3
Population: Intent-to-treat = All randomized subjects who underwent at least 1 study transfusion
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Mirasol | Control
Number analyzed (Participants) | 111 | 112
seconds
  Day 0 | 10.08 (3.11) | 10.07 (4.02)
  Day 1 | 10.19 (2.86) | 9.71 (3.33)
  Day 2 | 9.36 (2.20) | 9.62 (2.48)
  Day 3 | 9.53 (2.28) | 9.97 (3.03)

16. Secondary Outcome: Coagulation Parameter in Patients - Activated Partial Thromboplastin Time
Description: Activated partial thromboplastin time measure in study participants. Study participants may have received 1 or 2 blood product transfusions over 3 days while on study. These measurements were taken relative to the first transfusion only, for consistency.
Time Frame: Days 0, 1, 2, 3
Population: Intent-to-treat = All randomized subjects who underwent at least 1 study transfusion
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Mirasol | Control
Number analyzed (Participants) | 111 | 112
seconds
  Day 0 | 29.61 (9.12) | 29.12 (9.47)
  Day 1 | 29.89 (7.47) | 29.0 (10.25)
  Day 2 | 28.54 (6.64) | 27.89 (6.45)
  Day 3 | 28.60 (6.33) | 29.68 (7.73)

17. Secondary Outcome: Coagulation Parameter in Patients - International Normalized Ratio (INR)
Description: INR measure in study participants. Study participants may have received 1 or 2 blood product transfusions over 3 days while on study. These measurements were taken relative to the first transfusion only, for consistency.
Time Frame: Days 0, 1, 2, 3
Population: Intent-to-treat = All randomized subjects who underwent at least 1 study transfusion
Measure: Mean (Standard Deviation); unit: ratio
Arm/Group | Mirasol | Control
Number analyzed (Participants) | 111 | 112
ratio
  Day 0 | 1.05 (0.26) | 1.04 (0.33)
  Day 1 | 1.07 (0.25) | 1.02 (0.27)
  Day 2 | 0.99 (0.19) | 1.01 (0.20)
  Day 3 | 1.00 (0.19) | 1.04 (0.25)

ADVERSE EVENTS:
Time Frame: 28 days
Description: From the time of the initial transfusion through the 28-day Final Follow-up Visit
Arm/Group | Mirasol | Control
Serious Adverse Events (participants affected / at risk) | 13/111 | 9/112
Other Adverse Events (participants affected / at risk) | 33/111 | 37/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirasol (N=111) | Control (N=112)
Pericardial effusion (Cardiac disorders) | 1 (1) | 0 (0)
Ovarian cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Uraemic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Liver carcinoma ruptured (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 (1) | 1 (1)
Asthenia (General disorders) | 1 (1) | 0 (0)
Endometrial cancer metastatic (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Atypical pneumonia (Infections and infestations) | 1 (1) | 0 (0)
Nephrotic syndrome (Renal and urinary disorders) | 1 (1) | 0 (0)
Hypoglycaemia (Metabolism and nutrition disorders) | 1 (1) | 2 (2)
Hodgkin's disease (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Urinary tract infection (Infections and infestations) | 1 (1) | 0 (0)
Encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 1 (1) | 0 (0)
Hepatic encephalopathy (Nervous system disorders) | 1 (1) | 0 (0)
Malaria (Infections and infestations) | 1 (1) | 1 (1)
Pelvic abscess (Infections and infestations) | 1 (1) | 0 (0)
Hepatic failure (Hepatobiliary disorders) | 0 (0) | 1 (1)
Loss of consciousness (Nervous system disorders) | 0 (0) | 1 (1)
Circulatory collapse (Vascular disorders) | 0 (0) | 1 (1)
Hyperkalaemia (Metabolism and nutrition disorders) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 1 (1)
Enterocutaneous fistula (Gastrointestinal disorders) | 0 (0) | 1 (1)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pyelonephritis (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Mirasol (N=111) | Control (N=112)
Allergic transfusion reaction (Injury, poisoning and procedural complications) | 5 (5) | 9 (9)
Febrile nonhaemolytic transfusion reaction (Injury, poisoning and procedural complications) | 4 (4) | 5 (5)
Malaria (Infections and infestations) | 7 (7) | 5 (5)
Hypertension (Vascular disorders) | 5 (5) | 3 (3)
Headache (Nervous system disorders) | 3 (3) | 4 (4)
Hypokalaemia (Metabolism and nutrition disorders) | 4 (4) | 2 (2)
Pyrexia (General disorders) | 2 (2) | 3 (3)
Chills (General disorders) | 0 (0) | 2 (2)
Vomiting (Gastrointestinal disorders) | 1 (1) | 2 (2)
Gastritis (Gastrointestinal disorders) | 0 (0) | 2 (2)
Tachypnoea (Respiratory, thoracic and mediastinal disorders) | 2 (2) | 0 (0)

LIMITATIONS AND CAVEATS:
Necessary powering for the overall number of transfusions even though a smaller subgroup of non-parasitaemic patients receiving parasitaemic blood was the a-priori defined population to be assessed. Sufficient power was nevertheless maintained.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less